CLINICAL TRIAL: NCT02162160
Title: Microbiological Impact of a Cream and the Feeling of Softness and Freshness in the Intimate Area of Women
Brief Title: Microbiological Impact of an Intimate Cream and Its Suitability to Contribute to the Feeling of Softness and Freshness in the Intimate Area of Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Consultant, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KI DS 2013
Record Dates: First submitted 2013-11-21; First posted 2014-06-12 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Post Menopausal Dryness in the Intimate Area of Women
Keywords: probiotic; post-menopausal; atrophic vaginitis
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic creme (Experimental): Women receing probiotic creme
  Interventions: Device: probiotic creme
- placebo (Placebo Comparator): Women receiving a moisturizer
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: probiotic creme — Probiotic creme applied
  Other Names: Ellen AB
  Arms: Probiotic creme
Drug: Placebo — Creme without probiotics applied in same manner
  Arms: placebo

SUMMARY:
Generate more information on the use of the Probiotic Intimate Crème regarding feeling of dryness and freshness in the intimate area, as well as to evaluate the Lactobacillus flora and presence of coliform bacteria in respect to E. coli in the intimate area of women before use of the crème and at the end of a 10 days crème-usage (day 8-10), as well as 10 days after (9-11 days) finished crème-usage.

The hypothesis is that lactobacilli can survive in the intimate area of postmenopausal women with use of a probiotic creme.

DETAILED DESCRIPTION:
The rational for using probiotics is that the humans are colonized by a numbers of microorganisms from birth. These microorganisms are the natural flora of the human body. This bacterial ecology may be imbalanced due different circumstances: excessive hygiene, use of antibiotics or other drugs, use of alcohol, smoking, stress, diabetes and many other factors. The natural bacterial flora in the external part of the genital tract might be promoted by help of intimate products containing probiotics.

The study objectives Generate more information on the use of the Probiotic Intimate Crème regarding feeling of dryness and freshness in the intimate area, as well as to evaluate the Lactobacillus flora and presence of coliform bacteria in respect to E. coli in the intimate area of women before and at the end of a 10 days crème-usage (day 8-10), as well as 10 (9-11) days after finished crème-usage.

The primary endpoint of the study Presence of at least one LN bacteria strain in the intimate area of women in the intervention group compared to the intimate area of women in the control group at the end of a 10 days crème-usage (Day 8-10), as well as 10 (9-11) days after finished crème-usage. The primary endpint will be measured by bacterial Culture.

None-parametric statistical analyses.

Secondary endpoints Obtain information about the coliform bacteria flora in respect to E. coli flora in the external intimate area before and at the end of the 10 days crème-usage (Day 8-10), as well as 10 days after finished crème-usage (9-11 days after).

Obtain information about the subjective feeling of dryness and freshness in the intimate of women before and at the end of the 10 days crème-usage (Day 8-10), as well as 10 days after finished crème-usage (9-11 days after).

Only descriptive statistics.

Blinding The active and comparative test product will be filled into white tubes with identical appearance.

The study will be conducted with double-blind design when neither the personnel at the clinic and the participants knows which product they are submitted/received. The study will also be blinded for the laboratory personnel analyzing the samples.

Randomization procedure The women will be randomly assigned to active or comparative test products. Based on a computer-generated list, before start of the study, nine tubes containing Probiotic Intimate Crème (the active product) and 9 tubes containing Soothing crème (the control product) will be randomly assigned to a number between 1 to 18, and the tubes labeled with the numbers. The numbered but otherwise visually identical tubes will delivered to the clinic before start of the study.

During the first visit, the participants will receive a tube consecutively in numerical order, as they are included in the study, i.e. according to their participant number.

The computer-generated randomization list and the product labeling will be carried out by people who don't have direct contact with the study participants.

Sample collection

Vaginal samples:

The samples will be taken by rolling sterile swabs over the upper third part of the lateral vaginal wall.

Labial samples:

For labial sampling, on the left side of the vulva near the vaginal orifice, the labia minor and major will be held apart and a sterile swab will be gently rubbed back and forth five times during rotation. The labial examination area will be approximately 2 cm2.

The swabs will then be placed in a prepared transport medium and sent to laboratory for analyses.

6.12. Study outline

Visit 1:

1. Women visiting the clinic will be recruited to the study. After obtained information (Appendix 1) and signed informed consent the women will be clinically examined for any clinical symptoms of Candida vaginitis (ocular examination) and bacterial vaginosis (Amsel's criteria). The dryness of the mucus membranes will be also examined and the vaginal pH measured using a pH-stick.
2. Women fulfilling the inclusion criteria will be randomized to 10 days use of test product (Probiotic Intimate Crème) or control product (Soothing Cream, ACO); 2 times daily, every morning and evening at bed time.
3. The women will receive detailed instructions about how to use the study products.
4. They will also asked to return the empty tube or remaining product at the end of study (Visit 3)
5. The women will answer a questioner regarding their subjective feeling of dryness and freshness in their intimate are and rate their feeling on a ten-point scale.
6. Samples with sterile swabs will be collected from vagina, labia and perineum (Sample 1-L, Sample 1-V) and sent to an independent laboratory for analyses.

Visit 2:

1. The 8th-10th day of the intimate crème-usage period, the women will return to the clinic. The dryness of their mucus membranes will be clinically examined and the vaginal pH.
2. They will answer a questioner regarding their subjective feeling of dryness and freshness in their intimate are and rate their feeling on a on a ten-point scale. They will also answer questions regarding their purchase intentions and intentions to recommend the product to other women.
3. Vaginal and labial swabs will be collected (Sample 2-L, Sample 2-V) and send to an independent laboratory for analyses.

Visit 3:

1. 9-11 days after the 10 days crème-usage period, the women will return to the clinic. The dryness of their mucus membranes will be clinically examined and the vaginal pH measured.
2. They will answer a questioner regarding their subjective feeling of dryness and freshness in their intimate are and rate their feeling on a ten-point scale. They will also answer questions regarding their purchase intentions and intentions to recommend the product to other women.
3. Vaginal and labial swabs will be collected. (Sample 3-L, Sample 3-V) and sent to an independent laboratory for analyses.

During each visit, data will be recorded in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* healthy women 45-65 years old
* with subjective dryness in the intimate area
* postmenopausal with last menstruation more than or equal to 3 years prior to entering the study
* being willing to abstain sexual intercourse during the study period

Exclusion Criteria:

* yeast infection or bacterial vaginosis
* use of antibiotics or antifungals
* use of estrogen
* participation in Another study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Presence of at least one LN bacteria strain in the intimate area of women in the intervention group | the end of a 10 days crème-usage
  Bacterial Culture of LN bacterial strains

SECONDARY OUTCOMES:
Obtain information about the coliform bacteria flora in respect to E. coli flora in the external intimate area | at the end of creme usage and 10 days after finished crème-usage (9-11 days after).
  Measured by bacterial Culture and subtyping by PCR
subjective feeling of dryness and freshness in the intimate of women | the end of the 10 days crème-usage (Day 8-10) and 10 days after finished crème-usage (9-11 days after)
  Assessed through self adminstered questionnair with grading of feeling of dryness and freshness on a scale from 0 (no dryness and feeling fresh) to 5 (max dryness and absolutely not feeling fresh)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp Kallner, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of Obstetrics and Gynecology, Dnderyds Hospital, Stockholm, Sweden